CLINICAL TRIAL: NCT05689151
Title: Treating Atopic Dermatitis With Abrocitinib and Its Impact in Real Life: An Observational Cohort Study To Describe the Effectiveness of Abrocitinib in Patients With Moderate-to-Severe Atopic Dermatitis.
Brief Title: A Study to Learn About Abrocitinib in Adult Patients With Moderate to Severe Atopic Dermatitis.
Acronym: ADAIR
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7451096; ADAIR (Other: Alias Study Number)
Record Dates: First submitted 2023-01-09; First posted 2023-01-19 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: Atopic dermatitis; AD; Eczema; Abrocitinib; JAK inhibitors; France; Dermatitis; Atopic; Inflammatory disease; dermatology
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis | interventions — abrocitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Abrocitinib — Study Drug for Observational Data Collection

SUMMARY:
The purpose of this study is to learn about the safety and effects of Abrocitinib in the real-life clinical setting given for the treatment of moderate to severe atopic dermatitis. Atopic dermatitis, or AD, is a long-lasting disease that causes inflammation, redness, and irritation of the skin.

This study is seeking participant who are older than 18 years with moderate-to-severe chronic AD. Participants must have no underlying medical conditions that prevent them from taking Abrocitinib.

All participants in this study will receive Abrocitinib as a tablet once daily. They can take Abrocitinib and use medicated topical treatment for AD at the same time.

We will examine the experiences of patients receiving the study medicine. This will help us determine if the study medicine is safe and helps in treating AD.

Participants will take part in this study for 24 months. During this time, they will visit the study clinic about 5 times (about 1 time every 4 to 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age at inclusion.
* Patients with clinical diagnosis of moderate-to-severe chronic atopic dermatitis (also referred to as atopic eczema) at inclusion according to the investigator and eligible for abrocitinib according to its marketing approval.
* Patients that have been informed of the study procedures and have signed the consent.

Exclusion Criteria:

* Patients for whom abrocitinib is contraindicated.
* Patients unable to follow and respect the study procedures and judged inapt to respond to the questions required for the study due to linguistical, psychological, social, or geographical reasons.
* Patients not affiliated to the French social security system.
* Patients deprived of liberty, under guardianship, or unable to provide oral consent.
* Patients participating in a clinical study assessing a medicinal treatment (patients can participate in registries and observatories).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of moderate to severe atopic dermatitis for whom the dermatologist has decided to initiate a treatment with Abrocitinib
Sampling Method: Non-Probability Sample
Enrollment: 183 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with an Investigator's Global Assessment (IGA) score of clear (0) or almost clear (1) (on a 5- point scale) and a reduction from baseline of ≥2 points | 16 weeks

SECONDARY OUTCOMES:
Proportion of patients with an Investigator's Global Assessment (IGA) score of clear (0) or almost clear (1) (on a 5- point scale) and a reduction from baseline of ≥2 points | 12, 18 and 24 months
Change in Eczema Area and Severity Index (EASI) score from baseline | 16 weeks and at 12, 18, and 24 months
Proportion of patients with an EASI75 and EASI90 | at 16 weeks and at 12, 18, and 24 months
Time to Peak Pruritis-Numerical Rate Scale (PP-NRS) response (improvement of ≥2 points from baseline) | at 2, 16 weeks
PP-NRS (response improvement of ≥2 points or ≥4 points from baseline) | at 2, 16, 24 weeks and at 12 months
Absolute change from baseline in PP-NRS score | at 2, 16, and 24 weeks, and at 12 months
Absolute change from baseline Atopic Dermatitis Control Test (ADCT) score | at 16 and 24 weeks, and at 12, 18, and 24 months
Absolute changes from baseline score of Epworth sleepiness scale | at 2, 16, and 24 weeks, and at 12 months
Proportion of patients with ≤2 days per week of topical therapies applications, on average, in the last 4 weeks | at 24 weeks and at 12 months
Duration of Drug Therapy | Baseline to 24 months
Duration of each dosage | Baseline to 24 months
Proportion of patients with each regimen and changes over the treatment period | Baseline to 24 months
Proportion of patient with temporary treatment discontinuation | Baseline to 24 months
Proportion of patient with permanent treatment discontinuation with reason | Baseline up to 24 months
Proportion of Participants Receiving Subsequent Treatment | Baseline to 24 months
Number of Participants With Any Changes in Dosing | Baseline to 24 months
Proportion of patient with temporary treatment discontinuation with reason | Baseline to 24 months
Proportion of responders by items of Treatment Physician Satisfaction Questionnaire score (5-points Likert scale) | 16 and 24 weeks, and at 12 months
Demographic Characteristic of Participants: Age | Baseline
Demographical Characteristics of Participants:sex | Baseline
Demographic Characteristic of Participants: Body Mass Index | Baseline
Disease Characteristics of Participants: IGA score | Baseline
Disease Characteristics of Participants: EASI score | Baseline
Disease Characteristics of Participants: % of BSA involvement | Baseline
Disease Characteristics of Participants: PRO data | Baseline
Demographic Characteristics of Participants: history of treatment for atopic dermatitis | Baseline
Disease Characteristics of Participants: history of the disease | baseline
Demographic Characteristic of Participants: Comorbidities | Baseline
Hematological and lipid biological parameters | At baseline and 16 weeks
Proportion of patients with serious events | at 16 weeks, 12,18,24 months
Proportion of patients with non-serious adverse events | at 16 weeks, 12,18,24 months
Number of scratching episodes during the evening sleep period that occur pre treatment versus on treatment | At most 1 week before initiating abrocitinib and for 2 weeks on abrocitinib
  Data collection (scratch and sleep) from accelerometer monitor
Duration of time scratching during the evening sleep period that occur pre treatment versus on treatment | At most 1 week before initiating abrocitinib and for 2 weeks on abrocitinib
  Measure by accelerometer monitor
Compare change from pre-treatment to on-treatment measures of sleep quantity | At most 1 week before initiating abrocitinib and for 2 weeks on abrocitinib
  Measure by accelerometer monitor
Compare change from pre-treatment to on-treatment measures of Total sleep opportunity | At most 1 week before initiating abrocitinib and for 2 weeks on abrocitinib
  Measure by accelerometer monitor
Compare change from pre-treatment to on-treatment measures of Sleep efficiency | At most 1 week before initiating abrocitinib and for 2 weeks on abrocitinib
  Measure by accelerometer monitor
Compare change from pre-treatment to on-treatment measures of Total time asleep | At most 1 week before initiating abrocitinib and for 2 weeks on abrocitinib
  Measure by accelerometer monitor
Compare change from pre-treatment to on-treatment measures of Sleep onset latency | At most 1 week before initiating abrocitinib and for 2 weeks on abrocitinib
  Measure by accelerometer monitor
Compare change from pre-treatment to on-treatment measures of Wake after sleep onset and Number of wake bouts | At most 1 week before initiating abrocitinib and for 2 weeks on abrocitinib
  Measure by accelerometer monitor

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- France (30):
  - CHU Amiens-Picardie - Site Nord, Amiens, Somme
  - CHU Besancon - Hopital Jean Minjoz, Besançon
  - Polyclinique Reims Bezannes, Bezannes
  - Chu Bordeaux Hopital Saint Andre, Bordeaux
  - CHU Brest Hopital Morvan, Brest
  - CHU de Caen, Caen
  - Ch de Calais, Calais
  - Ch William Morey, Chalon-sur-Saône
  - CHU Clermont Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand
  - Chu Estaing, Clermont-Ferrand
  - Hopital Henri Mondor, Créteil
  - Chu Dijon, Dijon
  - Hopital Franco Britannique, Levallois-Perret
  - Hopital Claude Huriez, Lille
  - CH de Martigues, Martigues
  - CHU Montpellier, Montpellier
  - Hopital Emile Muller, Mulhouse
  - Hopital Hotel Dieu, Nantes
  - Hopital Cochin, Paris
  - Hopital Tenon, Paris
  - Hopital Saint Louis (APHP) - Service Hematologic Senior, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - Hopital Pontchaillou, Rennes
  - Ch de Romans Sur Isere, Romans-sur-Isère
  - Hopital Charles Nicolle, Rouen
  - Chi Poissy Saint Germain En Laye, Saint-Germain-en-Laye
  - Hopital Bégin, Saint-Mandé
  - Hopital Larrey, Toulouse
  - Ch de Valenciennes, Valenciennes
  - CHU Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451096